CLINICAL TRIAL: NCT07360457
Title: Association of GLP1 Analogues and SGLT2 Inhibitors With the Risk of Osteoarthritis in Type 2 Diabetic Patients
Brief Title: GLP1 Analogues and the Risk of Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Lecturer of clinical pharmacy, Beni-Suef University
Other Study IDs: GLP1
Record Dates: First submitted 2026-01-08; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis
Keywords: GLP-1
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium-Glucose Transporter 2 Inhibitors; Hypoglycemic Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SGLT2 Group: T2DM patients receiving SGLT2 inhibitors for at least 1 year added to their standard of care
  Interventions: Drug: SGLT2 inhibitor
- GLP1 Group: T2DM patients receiving GLP1 analogues for at least 1 year added to their standard of care
  Interventions: Drug: GLP-1 analog
- Control group: T2DM patients receiving only standard of care
  Interventions: Drug: Antidiabetic

INTERVENTIONS:
Drug: GLP-1 analog — glucagon like peptide analogues
  Other Names: GLP1 receptor agonist
  Groups: GLP1 Group
Drug: SGLT2 inhibitor — sodium glucose transporter-2 inhibitors
  Other Names: gliflozin
  Groups: SGLT2 Group
Drug: Antidiabetic — Standard of care
  Other Names: Control
  Groups: Control group

SUMMARY:
Assessing the effects of GLP1 RA Vs SGLT2 Inhibitors vs. Standard of care in joint pain, physical function, stiffness, and improving Quality of Life for patients with type 2 diabetes.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a multifactorial joint disease related to multiple inflammatory pathways which are triggered by mechanical and cellular stress, leading to increased production of pro-inflammatory mediators, reactive oxygen species, advanced glycation end products (AGEs). These mediators promote the release of proteolytic enzymes, which degrade the cartilage matrix. A recent study emphasized on the relation between metabolic syndrome and OA, considering metabolic dysregulation as a major factor in OA progression.

GLP-1 receptor agonists lower blood sugar by boosting glucose-dependent insulin release, reducing glucagon secretion, and slowing stomach emptying. GLP-1RA is present in both healthy and osteoarthritic cartilage, indicating a direct effect on chondrocytes. so it can decrease the accumulation of AGEs, which is the main cause of OA. It also reduces appetite, leading to weight loss which decreases the mechanical stress on joints. GLP downregulates proinflammatory cytokines (IL-6, TNF-a). also inhibits NF-κB pathway. which has a role in promoting osteoclast formation, so GLP plays a protective role in OA.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged above 50 years old with a previous diagnosis of T2DM according to ADA 2025, who have been on either SGLT2 inhibitors or GLP-1 analogs for at least one year.

Exclusion Criteria:

* individuals with Type 1 Diabetes Mellitus
* non-diabetic individuals
* those taking prandial insulin
* patients with arthritis without osteoarthritis,
* those taking other medications contraindicated with study medications,
* pregnant or breastfeeding females
* those allergic to active ingredients,
* those using corticosteroids, Autoimmune disease patients or patients receiving immunotherapies, monoclonal antibody targeting TNF-α or IL-6.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 T2DM patients will be admitted in each group Group 1 : T2DM patients receiving SGLT2 inhibitors for at least 1 year added to their standard of care Group 2: T2DM patients receiving GLP1 analogues for at least 1 year added to their standard of care Group 3: T2DM patients receiving only standard of care
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC score | at Day 1
  A validated, self-administered questionnaire used to assess pain, stiffness, and physical function

SECONDARY OUTCOMES:
VAS pain score | at Day 1
  numerical measure to assess pain

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Elsayed, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No